CLINICAL TRIAL: NCT06664385
Title: Effect of a Concurrent Physical Exercise Program on Quality of Life in Hemodialysis Patients: Uncontrolled Clinical Trial
Brief Title: Effect of a Concurrent Physical Exercise Program in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Julian Flores Moreno (Other)
Collaborators: Fabián Rojas Larios (Unknown); Israel Pérez Palafox (Unknown); Luis Antonio Bermudez Aceves (Unknown); Universidad de Colima (Other)
Responsible Party: Sponsor-Investigator, Pedro Julian Flores Moreno, Ph.D. in Science, Universidad de Colima
Organization: Universidad de Colima (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI 2024/1/CR/CL/SFIS/187
Record Dates: First submitted 2024-10-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Chronic Renal Insufficiency; Hemodialysis
Keywords: Hemodialysis; Functional Capacity; physical exercise; Quality of life
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: non controlled clinical trial
Masking Description: The masking consists of the investigator not performing the physical evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- concurrent physical exercise (Active Comparator): It consists of an exercise method that combines strength and endurance. It has a duration of 6 weeks divided into three stages, adaptation, development and maintenance. That for the intervention group and for the control group will only be performing aerobic physical exercise according to their physical tolerance.
  Interventions: Other: concurrent physical exercise

INTERVENTIONS:
Other: concurrent physical exercise — It consists of a periodization which consists of three moments adapted to the patient's needs distributed in 6 weeks and increasing the intensity gradually.

SUMMARY:
Concurrent physical exercise is the method of combining strength and endurance that can be worked with in one session or in an exercise program. Therefore, the researchers seek to implement it in patients suffering from chronic renal failure with hemodialysis therapy and see if concurrent physical exercise improves quality of life levels and at the same time see the response of physical fitness, body composition and biochemistry.

DETAILED DESCRIPTION:
Introduction: The performance of physical exercise has positive effects in terms of quality of life, but when it is not performed consistently it triggers a sedentary lifestyle, which is reflected in overweight and obesity, in addition to developing chronic noncommunicable diseases, propitiating chronic kidney disease, which although, hereditary and environmental factors are also present in this pathology and as the disease progresses, chronic renal failure develops. Objective: To analyze the effect of a concurrent physical exercise program on quality of life in patients with chronic renal failure undergoing hemodialysis. Methods: Uncontrolled clinical trial in which a concurrent physical exercise program will be carried out for 6 weeks, performing physical evaluations such as 6-minute walk and manual strength by dynamometer, application of SF-36 questionnaires, measurement of urea, glucose, creatinine and albumin, in addition to analyzing body composition by electrical bioimpedance.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are cared for at the State Hemodialysis Center.
* Receive hemodialysis treatment 3 times per week.
* Sign the informed consent form.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with a history of fracture at less than 2 months of evolution.
* Patients with any rheumatologic disease (lupus or rheumatoid arthritis).
* Prostrate patients.
* Amputee patients.
* Positive patients (HIV).
* Uncontrolled comorbidities.

Elimination.

* Patients who make their voluntary withdrawal from the project. Inability to engage in physical exercise.
* Death.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the level of quality of life with the SF-36 questionnaire, which ranges from 0 to 100 points, the higher the score, the higher the quality of life. | six weeks
  To analyze the quality of life of the patients and after the intervention to measure it again to see if the exercise has an impact on the levels of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro J Flores, Doctor of Medical Sciences, Study Chair — Universidad de Colima
Locations (1):
- Centro Estatal de Hemodialisis IMSS bienestar, Colima, Colima, Mexico

IPD SHARING:
Plan to Share IPD: Yes
the plan to share information with other researchers is through the publication of different articles that can be extracted from the research.
Supporting Information: Study Protocol, ICF
Time Frame: The information will be available as of August 2025.
Access Criteria: In order to have access to these data, other researchers must be performing the same methodological design, so there is no point in sharing it with a different study design.

REFERENCES:
- [Background] Molina-Robles E, Colomer-Codinachs M, Roquet-Bohils M, Chirveches-Perez E, Ortiz-Jurado P, Subirana-Casacuberta M. Effectiveness of an educational intervention and physical exercise on the functional capacity of patients on haemodialysis. Enferm Clin (Engl Ed). 2018 May-Jun;28(3):162-170. doi: 10.1016/j.enfcli.2017.12.003. Epub 2018 Mar 2. English, Spanish. PMID 29503041
- [Background] Segura-Orti E. [Exercise in haemodyalisis patients: a literature systematic review]. Nefrologia. 2010;30(2):236-46. doi: 10.3265/Nefrologia.pre2010.Jan.10229. Epub 2010 Jan 21. Spanish. PMID 20098466
- See also: Magazine containing extensive information on hemodialysis and physical exercise. — https://www.nefrologiaaldia.org